CLINICAL TRIAL: NCT03055338
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled Clinical Trial of the Efficacy and Safety of MK-8189 Using Risperidone as an Active Control in Subjects Experiencing an Acute Episode of Schizophrenia
Brief Title: An Active-Controlled Early Phase Study of MK-8189 in Adults With Schizophrenia (MK-8189-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8189-005; MK-8189-005 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Results first posted 2018-12-26 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia, Acute Episode
Keywords: Schizophrenia, acute episode; Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders
MeSH Terms: conditions — Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders | interventions — MK-8189; Risperidone

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups in parallel for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blind/masking technique will be used. MK-8189 and risperidone will be packaged identically relative to their respective matching placebo so that blinding/masking is maintained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MK-8189 (Experimental): Participants receive MK-8189 (4 mg controlled release [CR] oral tablet[s]) in combination with placebo matching risperidone (oral capsule[s]) once daily (QD) for 4 weeks. Over the initial 7 treatment days, MK-8189 is titrated from 4 mg to 12 mg as follows: 4 mg (1 tablet; Day 1); 8 mg (2 tablets; Day 4); and 12 mg (3 tablets; Day 7). Placebo matching risperidone is also titrated as follows: 1 capsule (Day 1), 2 capsules (Day 4), and 3 capsules (Day 7). After Day 7, MK-8189 is maintained at 12 mg (3 tablets) in combination with placebo matching risperidone (3 capsules), QD for 3 weeks.
  Interventions: Drug: MK-8189; Drug: Placebo matching risperidone
- Risperidone (Active Comparator): Participants receive risperidone (2 mg oral capsule[s]) in combination with placebo matching MK-8189 (oral tablet[s]), QD for 4 weeks. Over the initial 7 treatment days, risperidone is titrated from 2 mg to 6 mg as follows: 2 mg (1 capsule; Day 1); 4 mg (2 capsules; Day 4); and 6 mg (3 capsules; Day 7). Placebo matching MK-8189 is also titrated as follows: 1 tablet (Day 1), 2 tablets (Day 4), and 3 tablets (Day 7). After Day 7, risperidone is maintained at 6 mg (3 capsules) in combination with placebo matching MK-8189 (3 tablets), QD for 3 weeks.
  Interventions: Drug: Risperidone; Drug: Placebo matching MK-8189
- Placebo (Placebo Comparator): Participants receive both placebo matching MK-8189 (oral tablet[s]) as well as placebo matching Risperidone (oral capsule[s]), QD for 4 weeks. Over the initial 7 treatment days, placebo matching both MK-8189 and risperidone are respectively titrated as follows: 1 tablet/1 capsule (Day 1); 2 tablets/2 capsules (Day 4); and 3 tablets/3 capsules (Day 7). After Day 7, placebo matching both MK-8189 and risperidone are respectively maintained at 3 tablets/3 capsules, QD for 3 weeks.
  Interventions: Drug: Placebo matching MK-8189; Drug: Placebo matching risperidone

INTERVENTIONS:
Drug: MK-8189 — Oral CR tablets (4 mg) administered QD at the following dose strengths: 4 mg (1 tablet); 8 mg (2 tablets); 12 mg (3 tablets)
  Arms: MK-8189
Drug: Risperidone — Oral capsules (2 mg) administered QD at the following dose strengths: 2 mg (1 capsule); 4 mg (2 capsules); 6 mg (3 capsules)
  Arms: Risperidone
Drug: Placebo matching MK-8189 — Oral placebo tablet(s) matching the MK-8189 tablet, administered QD.
  Arms: Placebo; Risperidone
Drug: Placebo matching risperidone — Oral placebo capsule(s) matching the risperidone capsule, administered QD.
  Arms: MK-8189; Placebo

SUMMARY:
This will be a randomized, placebo-controlled, parallel-group, multi-site, double-blind trial of MK-8189 compared with placebo, using Risperidone as an active control. The participants will be adult subjects experiencing an acute episode of schizophrenia, according to the criteria specified in the Diagnostic and Statistical Manual of Mental Disorders, 5th ed. (DSM-5). This study will be up to 7 weeks in duration, with up to 7 site visits for each participant. The study will consist of a Screening/tapering period (up to one week long), a 4-week treatment period, and a 14-day follow-up period. The primary objective will be to assess symptoms of schizophrenia at 4 weeks, and to assess safety and tolerability during treatment and post-treatment follow-up. The secondary objective will be to assess the severity of schizophrenia at 4 weeks. The primary hypothesis is that MK-8189 is superior to placebo in reducing the overall symptoms of schizophrenia as assessed by the mean change from baseline in the Positive and Negative Syndrome Scale (PANSS) total score after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age at Screening
* Male
* Female not of reproductive potential (e.g., postmenopausal or has had a hysterectomy), or agrees to practice abstinence or use acceptable contraception
* Meets the diagnostic criteria for schizophrenia according to the DSM-5 criteria, or has a past diagnosis of schizophrenia with the onset of the first episode being >=1 year prior to study entry, and has illness duration of <=20 years
* Is confirmed to be experiencing an acute episode of schizophrenia
* Minimum PANSS score >= 80 at Screening
* Has a score of >=4 in 3 or more of the following items (delusions, conceptual disorganization, hallucinatory behavior, grandiosity, suspiciousness/persecution) in the positive subscale of the PANSS at Screening
* Has a CGI-S score >= 4 at Screening
* Is able to taper off psychotropic medications without significant destabilization or increased suicidality
* Has responded positively to an antipsychotic medication other than clozapine in a prior psychotic episode
* Has an identified responsible external contact person who has regular contact (no less than once per week) with the participant

Exclusion Criteria:

* Is currently under involuntary commitment because he/she is considered a danger to himself/herself or others
* Is unwilling to remain hospitalized for the duration of trial treatment
* Is currently participating in or has participated in an interventional clinical research study <=6 months prior to Screening, or has participated in more than one interventional clinical trial research study within 12 months prior to Screening
* Is unwilling to allow audio/video taping of the Mini International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorders (MINI) and/or PANSS interview at Screening and Baseline
* Is currently being treated with and benefiting from medications with a moderate or strong inhibiting or inducing effect on Cytochrome P450 (CYP) 3A and/or CYP2C9 and/or sensitive substrates of CYP2B6
* Has a history of malignancy <= 5 years except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Has a body mass index <18.5 or >40 kg/m˄2
* Has a history of treatment-resistant schizophrenia
* Has a prolactin laboratory value of >= 5 times the upper limit of normal at Screening
* Has a known history or clinical evidence of clinically significant hepatic, cardiovascular, or renal disease, or of untreated narrow-angle glaucoma- Has ever been diagnosed with epilepsy or had any seizure disorder beyond one childhood febrile seizure
* Has known serological evidence of human immunodeficiency virus (HIV) antibody
* Has a history of neuroleptic malignant syndrome
* Has a current diagnosis other than schizophrenia, or a comorbid diagnosis primarily responsible for current symptoms and functional impairment
* Has a known history of borderline personality disorder, antisocial personality disorder, or bipolar disorder
* Has a known history of traumatic brain injury, or Alzheimer's disease or another form of dementia
* Currently meets DSM-5 criteria for substance abuse or alcohol use disorder
* Is at imminent risk of self-harm or harm to others

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (28):
- United States (28):
  - Woodland International Research Group, LLC ( Site 0001), Little Rock, Arkansas
  - Woodland Research Northwest, LLC ( Site 0014), Rogers, Arkansas
  - CITRIALS ( Site 0013), Bellflower, California
  - Comprehensive Clinical Development ( Site 0049), Cerritos, California
  - Collaborative Neuroscience Network, LLC ( Site 0057), Garden Grove, California
  - Behavioral Research Specialists, LLC ( Site 0006), Glendale, California
  - Synergy East ( Site 0003), Lemon Grove, California
  - NRC Research Institute ( Site 0043), Orange, California
  - CNRI - Los Angeles, LLC ( Site 0026), Pico Rivera, California
  - Artemis Institute for Clinical Research ( Site 0027), San Diego, California
  - Schuster Medical Research Institute ( Site 0032), Sherman Oaks, California
  - Collaborative Neuroscience Network, LLC ( Site 0046), Torrance, California
  - Larkin Community Hospital Behavioral Health Services ( Site 0020), Hollywood, Florida
  - Clinical Research Centers of America, LLC ( Site 0038), Oakland Park, Florida
  - Aspire Health Partners ( Site 0016), Orlando, Florida
  - Radiant Research - Atlanta ( Site 0008), Atlanta, Georgia
  - Atlanta Center For Medical Research ( Site 0056), Atlanta, Georgia
  - Alexian Center for Psychiatric Research ( Site 0015), Hoffman Estates, Illinois
  - Lake Charles Clinical Trials, LLC ( Site 0040), Lake Charles, Louisiana
  - CBH Health, LLC ( Site 0022), Gaithersburg, Maryland
  - Precise Research Centers ( Site 0018), Flowood, Mississippi
  - Psych Care Consultants Research ( Site 0025), St Louis, Missouri
  - St. Louis Clinical Trials, LLC ( Site 0012), St Louis, Missouri
  - Altea Research Institute ( Site 0017), Las Vegas, Nevada
  - Radiant Research -CliniLabs ( Site 0037), New York, New York
  - Midwest Clinical Research Unit ( Site 0041), Dayton, Ohio
  - InSite Clinical Research ( Site 0033), DeSoto, Texas
  - Pillar Clinical Research, LLC ( Site 0004), Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mukai Y, Lupinacci R, Marder S, Snow-Adami L, Voss T, Smith SM, Egan MF. Effects of PDE10A inhibitor MK-8189 in people with an acute episode of schizophrenia: A randomized proof-of-concept clinical trial. Schizophr Res. 2024 Aug;270:37-43. doi: 10.1016/j.schres.2024.05.019. Epub 2024 Jun 8. PMID 38851166

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-8189: Participants receive MK-8189 (4 mg controlled release [CR] oral tablet[s]) in combination with placebo matching risperidone (oral capsule[s]) once daily (QD) for 4 weeks. Over the initial 7 treatment days, MK-8189 is titrated from 4 mg to 12 mg as follows: 4 mg (1 tablet; Day 1); 8 mg (2 tablets; Day 4); and 12 mg (3 tablets; Day 7). Placebo matching risperidone is mock titrated as follows: 1 capsule (Day 1), 2 capsules (Day 4), and 3 capsules (Day 7). After Day 7, MK-8189 is maintained at 12 mg (3 tablets) in combination with placebo matching risperidone (3 capsules), QD for 3 weeks.
- Risperidone: Participants receive risperidone (2 mg oral capsule[s]) in combination with placebo matching MK-8189 (oral tablet[s]), QD for 4 weeks. Over the initial 7 treatment days, risperidone is titrated from 2 mg to 6 mg as follows: 2 mg (1 capsule; Day 1); 4 mg (2 capsules; Day 4); and 6 mg (3 capsules; Day 7). Placebo matching MK-8189 is mock titrated as follows: 1 tablet (Day 1), 2 tablets (Day 4), and 3 tablets (Day 7). After Day 7, risperidone is maintained at 6 mg (3 capsules) in combination with placebo matching MK-8189 (3 tablets), QD for 3 weeks.
- Placebo: Participants receive both placebo matching MK-8189 (oral tablet[s]) as well as placebo matching Risperidone (oral capsule[s]), QD for 4 weeks. Over the initial 7 treatment days, placebo matching both MK-8189 and risperidone are respectively mock titrated as follows: 1 tablet/1 capsule (Day 1); 2 tablets/2 capsules (Day 4); and 3 tablets/3 capsules (Day 7). After Day 7, placebo matching both MK-8189 and risperidone are respectively maintained at 3 tablets/3 capsules, QD for 3 weeks.
Period: Overall Study
Arm/Group | MK-8189 | Risperidone | Placebo
Started | 90 | 45 | 89
Completed | 72 | 34 | 77
Not Completed | 18 | 11 | 12
Not completed — Lost to Follow-up | 9 | 2 | 3
Not completed — No Post-treatment Protocol Contact | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Withdrawal by Subject | 9 | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- MK-8189: Participants receive MK-8189 (4 mg CR oral tablet[s]) in combination with placebo matching risperidone (oral capsule[s]) QD for 4 weeks. Over the initial 7 treatment days, MK-8189 is titrated from 4 mg to 12 mg as follows: 4 mg (1 tablet; Day 1); 8 mg (2 tablets; Day 4); and 12 mg (3 tablets; Day 7). Placebo matching risperidone is mock titrated as follows: 1 capsule (Day 1), 2 capsules (Day 4), and 3 capsules (Day 7). After Day 7, MK-8189 is maintained at 12 mg (3 tablets) in combination with placebo matching risperidone (3 capsules), QD for 3 weeks.
- Total: Total of all reporting groups
Arm/Group | MK-8189 | Risperidone | Placebo | Total
Number analyzed (Participants) | 90 | 45 | 89 | 224
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.4 (7.4) | 37.3 (8.0) | 35.6 (7.6) | 37.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 8 | 17 | 48
  Male | 67 | 37 | 72 | 176
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 65 | 37 | 65 | 167
  White | 21 | 8 | 20 | 49
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Positive and Negative Syndrome Scale (PANSS) Total Score [Mean (Standard Deviation); unit: Score on a Scale] — The PANSS assesses the severity of schizophrenia symptoms through a clinician-rated inventory of 30 items organized in 3 subscales: 1) positive subscale (7 items); 2) negative subscale (7 items); and 3) general psychopathology subscale (16 items). For each item, symptoms are scored from 1 (absent) to 7 (extreme) and sum to a total PANSS score (range: 30-210). Higher scores reflect more severe symptoms of schizophrenia. Population: Includes all randomized participants who: 1) received ≥1 dose of study treatment; 2) had a baseline PANSS assessment; and 3) had ≥1 post-randomization observation for PANSS score subsequent to ≥1 dose of study treatment.
  Score on a Scale
    number analyzed (Participants) | 89 | 40 | 89 | 218
    (all) | 95.1 (10.4) | 95.3 (12.4) | 96.2 (9.6) | 95.6 (10.45)
Clinical Global Impression Severity of Illness (CGI-S) Score [Mean (Standard Deviation); unit: Score on a Scale] — The CGI-S is a 7-point clinician-rated scale for assessing the global severity of the participant's illness. Possible CGI-S scores range from 1 (participant normal, not ill) to 7 (participant extremely ill). Population: Includes all randomized participants who: 1) received ≥1 dose of study treatment; 2) had a baseline CGI-S assessment; and 3) had ≥1 post-randomization observation for CGI-S score subsequent to ≥1 dose of study treatment.
  Score on a Scale
    number analyzed (Participants) | 89 | 40 | 89 | 218
    (all) | 4.9 (0.6) | 5.0 (0.7) | 5.0 (0.4) | 4.9 (0.57)
Duration of Illness [Count of Participants; unit: Participants]
  <= 10 Years | 31 | 18 | 32 | 81
  > 10 Years | 59 | 27 | 57 | 143

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean (LSM) Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at Week 4
Description: The LSM change from baseline at week 4 was assessed for PANSS total score. The PANSS assesses the severity of schizophrenia symptoms through a clinician-rated inventory of 30 items organized in 3 subscales: 1) positive subscale (7 items); 2) negative subscale (7 items); and 3) general psychopathology subscale (16 items). For each item, symptoms are scored from 1 (absent) to 7 (extreme) and sum to a total PANSS score (range: 30-210). Higher scores reflect more severe symptoms of schizophrenia. Further, reduced symptom severity over time is reflected by decreases in score.
Time Frame: Baseline and Week 4
Population: Includes all randomized participants who: 1) received ≥1 dose of study treatment; 2) had a baseline PANSS assessment; and 3) had ≥1 post-randomization observation for PANSS score subsequent to ≥1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-8189 | Risperidone | Placebo
Number analyzed (Participants) | 89 | 40 | 89
Score on a Scale | -14.6 [-18.2 to -11.1] | -17.2 [-22.8 to -11.6] | -10.0 [-13.7 to -6.2]
Statistical Analysis 1: Comparison: MK-8189 vs Risperidone; Test type: Superiority; p = 0.440, Longitudinal ANCOVA; Includes terms for treatment, baseline PANSS total score, age, duration of illness, week, and the interaction of week by treatment; Difference in LSM = 2.6, 95% CI 2-sided [-4.0 to 9.2] — Difference in LSM = MK-8189 - Risperidone
Statistical Analysis 2: Comparison: MK-8189 vs Placebo; Test type: Superiority; p = 0.074, Longitudinal ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in LSM = -4.7, 95% CI 2-sided [-9.8 to 0.5] — Difference in LSM = MK-8189 - Placebo
Statistical Analysis 3: Comparison: Risperidone vs Placebo; Test type: Superiority; p = 0.033, Longitudinal ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in LSM = -7.3, 95% CI 2-sided [-14.0 to -0.6] — Difference in LSM = Risperidone - Placebo

2. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE)
Description: The percentage of participants experiencing an AE was assessed. An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 6 weeks
Population: Includes all randomized and treated participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-8189 | Risperidone | Placebo
Number analyzed (Participants) | 90 | 45 | 89
Percentage of Participants | 71.1 | 77.8 | 53.9
Statistical Analysis 1: Comparison: MK-8189 vs Placebo; Test type: Other; Difference in % versus Placebo = 17.2, 95% CI 2-sided [3.0 to 30.8] — Difference in % = MK-8918 - Placebo; Based on Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an Adverse Event
Description: The percentage of participants discontinuing study treatment due to an AE was assessed. An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 4 weeks
Population: Includes all randomized and treated participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-8189 | Risperidone | Placebo
Number analyzed (Participants) | 90 | 45 | 89
Percentage of Participants | 6.7 | 8.9 | 7.9
Statistical Analysis 1: Comparison: MK-8189 vs Placebo; Test type: Other; Difference in % versus Placebo = -1.2, 95% CI 2-sided [-9.6 to 7.0] — Difference in % = MK-8918 - Placebo; Based on Miettinen & Nurminen method

4. Secondary Outcome: Least Squares Mean (LSM) Change From Baseline in the Clinical Global Impression-Severity of Illness (CGI-S) Score at Week 4
Description: The LSM change from baseline at week 4 was assessed for CGI-S score. The CGI-S is a 7-point clinician-rated scale for assessing the global severity of the participant's illness. Possible CGI-S scores range from 1 (participant normal, not ill) to 7 (participant extremely ill). Further, a decrease in CGI-S score indicates reduced severity of the participant's illness.
Time Frame: Baseline and Week 4
Population: Includes all randomized participants who: 1) received ≥1 dose of study treatment; 2) had a baseline CGI-S assessment; and 3) had ≥1 post-randomization observation for CGI-S score subsequent to ≥1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-8189 | Risperidone | Placebo
Number analyzed (Participants) | 89 | 40 | 89
Score on a Scale | -0.9 [-1.1 to -0.6] | -1.0 [-1.4 to -0.7] | -0.7 [-0.9 to -0.4]
Statistical Analysis 1: Comparison: MK-8189 vs Risperidone; Test type: Other; Difference in LSM = 0.2, 95% CI 2-sided [-0.2 to 0.6] — Difference in LSM = MK-8189 - Risperidone
Statistical Analysis 2: Comparison: MK-8189 vs Placebo; Test type: Other; Difference in LSM = -0.2, 95% CI 2-sided [-0.5 to 0.2] — Difference in LSM = MK-8189 - Placebo
Statistical Analysis 3: Comparison: Risperidone vs Placebo; Test type: Other; Difference in LSM = -0.4, 95% CI 2-sided [-0.8 to 0.1] — Difference in LSM = Risperidone - Placebo

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: The analysis population includes all randomized and treated participants.
Arm/Group | MK-8189 | Risperidone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/45 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/90 | 3/45 | 3/89
Other Adverse Events (participants affected / at risk) | 53/90 | 27/45 | 31/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8189 (N=90) | Risperidone (N=45) | Placebo (N=89)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Schizophrenia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8189 (N=90) | Risperidone (N=45) | Placebo (N=89)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 3 (3) | 5 (6)
Nausea (Gastrointestinal disorders) | 14 (15) | 4 (4) | 5 (5)
Vomiting (Gastrointestinal disorders) | 7 (7) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (4) | 2 (2)
Weight increased (Investigations) | 2 (2) | 8 (8) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 2 (2)
Akathisia (Nervous system disorders) | 16 (16) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 3 (4) | 4 (4) | 1 (1)
Dystonia (Nervous system disorders) | 8 (10) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 14 (18) | 5 (6) | 12 (17)
Lethargy (Nervous system disorders) | 1 (1) | 3 (6) | 1 (1)
Sedation (Nervous system disorders) | 7 (7) | 6 (6) | 2 (2)
Somnolence (Nervous system disorders) | 6 (6) | 2 (2) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1) | 3 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 7 (7) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT03055338/Prot_SAP_000.pdf